CLINICAL TRIAL: NCT01755377
Title: Evolution of Serologic Biomarkers and Diastolic Function and Segmentary Contractility Determined by Echocardiography After Treatment in Chagas Diseases
Brief Title: New Tools for the Diagnosis, Prognosis and Treatment Follow-up in Chagas Disease
Acronym: BIOMARCHA
Status: Completed | Type: Observational
Sponsor: Barcelona Centre for International Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMARCHA
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Chagas Disease: Participants with no Chagas Disease will be evaluated as a Control Group
- Chagas Disease: Participants diagnosed with Chagas Disease will be followed-up as a Case Group
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: Benznidazole
  Groups: Chagas Disease

SUMMARY:
Chagas disease is endemic to Latin America, and is of emerging importance in non-endemic countries because migration of people infected with T. cruzi. Current methods for diagnosis of T. cruzi infection are not ideal. Existing drugs for treatment are very limited, produce severe side-effects, and their effectiveness cannot be properly evaluated. Reliable biomarkers for prognosis, early diagnosis and effectiveness of treatment will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients from endemic areas (Latin America)
* Older than 18 years old and younger than 50
* With serological confirmation of Chagas Disease infection with two different techniques
* Indeterminate or initial cardiac form
* No previously treated for Chagas Disease

Exclusion Criteria:

* Co-morbidity: previous cardiac disease from other aetiology (ischemic, alcoholic or hypertensive), active inflammatory or immunology diseases for another agent. Hepatic disfunction
* Pregnancy or lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Migrants from Latin America visiting the Tropical Medicin Clinic
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Biomarkers for prognosis, early diagnosis and effectiveness of treatment. | 2 years
  * Conventional polymerase chain reaction of T. cruzi in blood
  * Measurement of Brain natriuretic factor
  * Measurement of Prothrombotic factors
  * Measurement of antibodies against specific proteins of the trypomastigote of T. cruzi
  * Investigation of the phylogenetics of the parasite and the role of the lineages of T.cruzi in the clinical presentation and disease's progression

SECONDARY OUTCOMES:
Cardiac function after antiparasitic treatment | 2 years
  - Correlation between biomarkers and alterations of the left ventricle diastolic function and segmentary contractility after antiparasitic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Gascón, PhD, Principal Investigator — Barcelona Centre for International Health Research (CRESIB)
Locations (1):
- International Health Department, Hospital Clinic, Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Aldasoro E, Posada E, Requena-Mendez A, Calvo-Cano A, Serret N, Casellas A, Sanz S, Soy D, Pinazo MJ, Gascon J. What to expect and when: benznidazole toxicity in chronic Chagas' disease treatment. J Antimicrob Chemother. 2018 Apr 1;73(4):1060-1067. doi: 10.1093/jac/dkx516. PMID 29351667